CLINICAL TRIAL: NCT04028791
Title: Metabolic and Vascular Response to Exercise in Sickle Cell Trait Carriers: Effect of Hot Environment
Brief Title: Sickle Cell Trait and Exercise, Effect of Hot Environment
Acronym: TDex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the French West Indies and French Guiana (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Sophie Antoine-Jonville, Director, University of the French West Indies and French Guiana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017-A02226-47
Record Dates: First submitted 2019-07-16; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Sickle Cell Trait; Environmental Exposure; Adverse Effect
Keywords: Exercise, sickling, rhamdomyolysis, oxidative stress
MeSH Terms: conditions — Sickle Cell Trait; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants in each group (AA, AS) will carry out the following 3 sessions:
  1. Exercise performed in hot environment (33 °C) with recovery in the same environment
  2. Exercise and recovery performed in a control (thermoneutral) environment (22 °C),
  3. Exercise performed in a hot environment (33 °C) with recovery in a thermoneutral, environment (22 °C).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AS and AA (Experimental): Participants will be submitted to 45 minutes of exercise on ergocycle.
  Interventions: Other: Exercise on ergocycle

INTERVENTIONS:
Other: Exercise on ergocycle — The exercise includes 15 minutes of warm up, then participants will be asked to pedal as fast as possible for 6 seconds. The test of 6 seconds will be repeated twice or more with recovery each time

SUMMARY:
The heterozygous form of sickle cell disease is clinically asymptomatic. Nevertheless, it was observed that, the sickle cell trait is associated with serious medical complications especially during intense physical efforts. Moreover, the exposure to a hot environment (tropical climate) is suspected to be a determining factor in the occurrence of these medical complications.

However, the relationship between sickle cell trait and death during effort is not well established. Furthermore, the cascade of events that usually cause sickle cell crisis such as red blood cells sickling and rhabdomyolysis and which affect microcirculation are not known.

Our main objective in this study is to verify whether young healthy active men with sickle cell trait have reactive hyperemia to their hemoglobinemic condition during exercise; to identify the contribution of hot environment on these possible disturbances; and to determine underlying mechanisms.

In addition, disturbances in the regulation of glucose metabolism in healthy subjects under hot environment have been reported, marked by a significant increase in postprandial blood glucose. Therefore, this project is also intended to assess the contribution of the disturbance of glycoregulation during exercise under hot environment in active sickle cell trait carriers. The imbalance of pro and anti oxidant agents, the adhesion and inflammation markers will also be evaluated.

Results of this study will allow a better understanding of physio-pathological mechanisms leading to vascular accidents during exercise under tropical climate in young healthy sickle cell trait carriers; and to identify physical activity programs and nutritional interventions adapted to patients with sickle cell disease under hot environment.

DETAILED DESCRIPTION:
Introduction

The sickle cell disease is an inherited disorder characterized by abnormal hemoglobin called hemoglobin S or sickle hemoglobin in red blood cells of subjects. The homozygous form (hemoglobin SS) causes sickle cell anemia and is the most severe kind of sickle cell disease. Hemoglobin SC disease and hemoglobin Sβ thalassemia are two other common forms of sickle cell disease. The sickle cell trait carriers are person who inherited the hemoglobin S from one parent and a normal hemoglobin A from the other (heterozygous AS). These people are generally healthy. However, more and more cases of serious complications have been reported, especially during efforts and stays at high altitude like hemorheological and microcirculatory disturbances, and rhabdomyolysis. Increased percentage of red cell sicking was observed in sickle cell trait (AS) carriers compared to normal individual after 45 min of walking at 33°C of temperature. AS individuals also showed an impairment in red blood deformability at rest, at the end, and 24 hours after maximal exercise as compared to normal individuals AA, showing the vulnerability of red blood cells of these seemingly healthy subjects. The stiffness of red blood cells along with blood viscosity also increased in AS group compared to AA group, as consequence the risk of vascular accidents increases. In athletes and military warfighters, an exercise collapse and sudden death associated with sickle cell trait has been observed. Several cases of sudden death in AS individuals have been reported by many authors during exercise, however the exact causes remain very poorly understood.

As constraints related to exercise in tropical climate, it was observed a reduction of power and volemia due to dehydration, diversion of blood volume to the cutaneous territories. It was also reported an impairment of carbohydrate metabolism.

Our objectives in this work are:

* To characterize the microvascular response to exercise in a hot environment in sickle cell trait active young adults,
* To highlight biological mechanisms underlying any microvascular response specificities of the sickle cell trait carriers,
* To describe the vascular consequences of postprandial metabolic disturbances induced by exercise in hot environment,
* To understand fasting and post-prandial glucose metabolism at rest, during and after exercise,
* To test the recovery in a neutral thermal environment (22 °C) as a means of normalizing post-exercise vascular function.

Experimental protocol

Thirty male volunteers (15 healthy: AA and 15 sickle cell trait carriers: AS) non-smoking, aged 18-30 years, BMI between 19 and 25kg/m2 living in the Caribbean for at least 6 months will be enrolled in the study. All subjects will be in good health physically active (≥ 3h/week) with no history of heat stroke during exercise. They are not taking any medications and are not regularly consume alcohol.

Participants will be subjected to four experimental sessions:

1. A familiarization session at fasting in a warm environment (33 °C) in which resting parameters like reactive hyperemia index, tympanic temperature, heart rate, cerebral and muscular oxygenation, pulse wave velocity and electrocardiogram (ECG) will be measured. Then a test of the intensity of exercise (VO2max) will be performed followed by a medical interview.

   The other 3 sessions will be performed early in the morning at fasting with 45 minutes of exercise on ergocycle. The exercise includes 15 minutes of warm up, then participants will be asked to pedal as fast as possible for 6 seconds. The test of 6 seconds will be repeated twice or more with recovery each time. During exercise, hydration will be controlled (2.5 ml water / kg every 15 minutes), oxygen consumption will be measured; and microvascular function and blood samples taken at different times of experiment in each session (T0, T60, T75, T90, T120). The design of this study is a crossover trial divided into 3 sessions presented in randomized order:
2. Exercise performed in hot environment (33 °C) with recovery in the same environment.
3. Exercise and recovery performed in a control (thermoneutral) environment (22 °C)
4. Exercise performed in a hot environment (33 °C) with recovery in a thermoneutral environment (22 °C).

At the end of each session, a standardized meal will be given to each participant.

This study will be conducted in accordance with the guidelines developed in the Declaration of Helsinki, and all procedures were approved by the Committee for the Protection of Persons East-III. Written informed consent will be obtained from all participants.

Biochemical procedures

Blood samples will be use for hemorheological tests (viscosity of blood, stiffness, aggregability and sickling of red cells etc.) Dosage of creatine kinase (CK-MM, MB), myoglobin and troponin will be performed to assess the degree of rhabdomyolysis and the integrity of heart.

Glycemia and lactatemia will be determined using strips. Cortisol, insulin, adrenalin, glucagon and lactate dehydrogenase (LDH) assays will be performed using appropriated kits.

Plasma inflammatory profile will be determined by measuring markers such as myeloperoxidase (MPO), malondialdehyde (MDA), advanced oxidation protein products (AOPP), nitrotyrosin, and endothelin-1 using appropriated kits.

Adhesion molecules such as VCAM-1, ICAM-1 and P-selectin will be measured using ELISA kit from Diaclone or Eurobio.

The oxidative stress on red blood cells will be assessed by measuring glutathione ratio GSSH/GSSG, superoxide dismutase (SOD), catalase, and glutathione peroxidase (GPx).

Statistical analysis Data will be expressed as means with their standard errors. Statistical analyses will be performed with SPSS for MAC and p < 0·05 considered statistically signiﬁcant.

All the data will be analysed by using repeated-measures ANOVA followed by Post hoc comparisons with the Student's paired t test. The tests of Kolmogorov-Smirnov, Newman Keuls and Duncan will be applied as appropriate.

Expected outcomes

* Better understanding of physio-pathological mechanisms leading to severe vascular events following physical exercise in tropical climate in healthy sickle cell carriers.
* Opening of tracks for identification of physical activity programs and nutritional interventions adapted to sickle cell patients in hot environment.
* Understanding of mechanisms leading to disturbances of glucose metabolism under tropical climate in AA and in AS subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 25kg/m2,
* Be living in the Caribbean for at least 6 months health
* Be physically active (≥ 1350 METs/week)
* No history of heat stroke during exercise
* No taking any medications
* Not regularly consuming alcohol
* Have the ability and willingness to issue consent written, free and enlightened

Exclusion Criteria:

* Have any other hemoglobinemic status than AA or AS.
* Weight gain or loss of more than 2 kg in the last 6 month.
* Food allergy to any of ingredients coming into the composition of test meals or that may result from a cross-contamination during manufacture: eggs and eggs products, gluten, milk and milk-based products (including lactose), soybean and soy products, fruit hulls (almonds, hazelnuts, walnuts, cashew nuts, pecan, macadamia, Brazil, Queensland, pistachios) and products made of these fruits.
* Monitoring a particular diet
* Any chronic metabolic pathology, cardiovascular, neurovascular, renal, respiratory, neuromuscular, musculoskeletal or articular known
* Any disorder of the ear (infections, tumors, perforated eardrums, polyps)
* Any infectious disease or inflammatory and infectious condition

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Microvascular function | 2 hours
  Reactive hyperemia index (arbitrary units) will be assessed at rest, during exercise and during recovery in hot and thermoneutral environment

SECONDARY OUTCOMES:
Oxidative stress | 3 months
  Glutathione ratio GSSH/GSSG
Inflammation | 3 months
  Myeloperoxidase (MPO)
Adhesion molecules | 3 mois
  VCAM-1
Hemorheology | 24 hours
  hematocrit
Rhamdomyolysis | 3 months
  Creatine kinase
Oxydative stress marker | 3 months
  superoxide dismutase (SOD)

OTHER OUTCOMES:
Glucose metabolism | 3 months
  glucose

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Henri, Dr, Principal Investigator — Laboratoire ACTES, EA 3596 UFR STAPS, University of the French West Indies and French Guiana; Olivier Hue, PhD, Study Director — Laboratoire ACTES, EA 3596 UFR STAPS, University of the French West Indies and French Guiana; Mona Hedreville, Dr, Principal Investigator — Unités Urgences cardiologiques CHU, Pointe-à-Pitre/Abymes 97159
Locations (1):
- ACTES laboratory, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided
All autors have to discuss together before to decide

REFERENCES:
- [Background] Bergeron MF, Cannon JG, Hall EL, Kutlar A. Erythrocyte sickling during exercise and thermal stress. Clin J Sport Med. 2004 Nov;14(6):354-6. doi: 10.1097/00042752-200411000-00005. PMID 15523207
- [Background] Connes P, Sara F, Hardy-Dessources MD, Marlin L, Etienne F, Larifla L, Saint-Martin C, Hue O. Effects of short supramaximal exercise on hemorheology in sickle cell trait carriers. Eur J Appl Physiol. 2006 May;97(2):143-50. doi: 10.1007/s00421-006-0155-3. Epub 2006 Feb 28. PMID 16506056
- [Background] Faure C, Charlot K, Henri S, Hardy-Dessources MD, Hue O, Antoine-Jonville S. Impaired glucose tolerance after brief heat exposure: a randomized crossover study in healthy young men. Clin Sci (Lond). 2016 Jun 1;130(12):1017-25. doi: 10.1042/CS20150461. Epub 2016 Mar 15. PMID 26980346
- [Background] Kark JA, Posey DM, Schumacher HR, Ruehle CJ. Sickle-cell trait as a risk factor for sudden death in physical training. N Engl J Med. 1987 Sep 24;317(13):781-7. doi: 10.1056/NEJM198709243171301. PMID 3627196
- [Background] Kerle KK, Nishimura KD. Exertional collapse and sudden death associated with sickle cell trait. Mil Med. 1996 Dec;161(12):766-7. PMID 8990839
- [Background] Kerle KK, Runkle GP. Sickle cell trait and sudden death in athletes. JAMA. 1996 Nov 13;276(18):1472. No abstract available. PMID 8903257
- [Background] Le Gallais D, Bile A, Mercier J, Paschel M, Tonellot JL, Dauverchain J. Exercise-induced death in sickle cell trait: role of aging, training, and deconditioning. Med Sci Sports Exerc. 1996 May;28(5):541-4. doi: 10.1097/00005768-199605000-00001. PMID 9148081
- [Background] Monchanin G, Connes P, Wouassi D, Francina A, Djoda B, Banga PE, Owona FX, Thiriet P, Massarelli R, Martin C. Hemorheology, sickle cell trait, and alpha-thalassemia in athletes: effects of exercise. Med Sci Sports Exerc. 2005 Jul;37(7):1086-92. doi: 10.1249/01.mss.0000170128.78432.96. PMID 16015123
- [Background] O'Connor FG, Bergeron MF, Cantrell J, Connes P, Harmon KG, Ivy E, Kark J, Klossner D, Lisman P, Meyers BK, O'Brien K, Ohene-Frempong K, Thompson AA, Whitehead J, Deuster PA. ACSM and CHAMP summit on sickle cell trait: mitigating risks for warfighters and athletes. Med Sci Sports Exerc. 2012 Nov;44(11):2045-56. doi: 10.1249/MSS.0b013e31826851c2. PMID 22811029
- [Background] Quattrone RD, Eichner ER, Beutler A, Adams WB, O'Connor FG. Exercise collapse associated with sickle cell trait (ECAST): case report and literature review. Curr Sports Med Rep. 2015 Mar-Apr;14(2):110-6. doi: 10.1249/JSR.0000000000000137. PMID 25757006
- [Background] Wirthwein DP, Spotswood SD, Barnard JJ, Prahlow JA. Death due to microvascular occlusion in sickle-cell trait following physical exertion. J Forensic Sci. 2001 Mar;46(2):399-401. PMID 11305451